CLINICAL TRIAL: NCT04203849
Title: Prospective Cohort Study for Identifying Factors Predicting Clinical Outcomes of Breast Cancer Patients Treated With Radiotherapy
Brief Title: Prospective Cohort Study of Breast Cancer Patients Treated With Radiotherapy
Status: Enrolling by invitation | Type: Observational
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Tae Hyun Kim, Principal Investigator, National Cancer Center, Korea
Other Study IDs: NCC2019-0142
Record Dates: First submitted 2019-11-28; First posted 2019-12-18 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
breast cancer occurred 19,219cases in 2015 and is the second most common cancer among female cancers in the country. despite there's been a disease understanding and treatment developing through study, the prevalence and mortality of breast cancer have increased steadily over the last 15 years. In the last 20 years, through random clinical studies of breast cancer, radiation therapy is well-established standard therapy as postoperative supplement of invasive breast cancer and intraepithelial carcinoma but, the need for further study with new questions about radiation therapy has been raised through these studies. according to the prospective study outcome, the radiation treatment of the regional lymph node in breast cancer patients with lymph node positive increases the free-disease survival rate, radiation therapy for regional lymph node is being actively treated than in the past. on the contrary, the results of another study are being reported that treating regional lymph node may increase the risk of arm edema, radiation pneumonia and heart toxicity. In the recently, due to advancement in radiation therapy technique, the implement of new radiation therapy such as IMRT that reducing radiation dose to normal tissues of the axillary, lungs, heart and others has been actively attempted.

additional research is needed on dose-fractionation schedule, regional lymph node treatment, post-treatment toxicity of radiation therapy in breast cancer. this study establishes a prospective cohort at breast cancer patients with radiation treatment and analyze the local and regional lymph node control, recurrence, toxicity, radiation planning, clinical data, discover the factors that predict local control, regional control, overall survival, recurrence-free survival, toxicity for treatment, so we intend to construct basic data that establishes a radiation treatment strategy based on comprehensive outcomes and predictors.

ELIGIBILITY:
Inclusion Criteria:

* scheduled to be a radiotherapy at National cancer center
* agreed to participate in the study

Exclusion Criteria:

- disagreed to participate in the study

Min Age: 20 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: breast cancer patient
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2019-07-03 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2034-06-30 (Estimated)

PRIMARY OUTCOMES:
local and regional lymphnode control, free-recurrence, survival period | up to 6 month
  local and regional lymphnode control, free-recurrence, survival period is defined as the date of occurrence or end based of an event on the date of breast cancer diagnosis. the date of occurrence of an event means the progress of local and region lymph node by disease, the recurrence(or progression) of disease or the confirmed date of death and the date of disconnection means the final date on which the event was determined not to have occurred.
  * In follow up loss, the date on which survival is confirmed before follow up loss is disconnection date.
  * a cancer diagnosis date is calculated based on the date of radiological examination of the findings.

SECONDARY OUTCOMES:
therapeutic responses according to image examination | up to 6 month
  therapeutic responses according to image examination is calculated as the fraction of the subjects who showed either 'CR' or 'PR' according to the RECIST criteria.
  *Response Criteria (RECIST)
  * [Complete Response (CR)]: disappearance of all extranodal target lesion.
  * [Partial Response (PR)]: At least a 30% decrease in the SLD of target lesions, taking as reference the baseline sum diameters
  * [Stable Disease (SD)]: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD
  * [Progressive Disease (PD)]: SLD increased by at least 20% from the smallest value on study or a new tumor has been created.
toxicity of radiotherapy | up to 6 month
  toxicity is calculated as the fraction of toxicity higher than grade 3 according to CTCAE.

CONTACTS AND LOCATIONS:
Overall Officials: Tae H Kim, Ph.D, Principal Investigator — National Cancer Center, Korea
Locations (1):
- National Cancer Center Korea, Goyang-si, Gyeonggi-do, South Korea